CLINICAL TRIAL: NCT00951860
Title: Assessment of Autonomic Maturation in Neonatal Period and Early Neural Development From a Longitudinal Prospective Cohort : the AuBE Study
Brief Title: Assessment of Autonomic Maturation in Neonatal Period and Early Neural Development From a Longitudinal Prospective Cohort
Acronym: AUBE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0908020; 2009-A00325-52 (Other: AFSSAPS)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Fullterm Birth; Neonate; Prematurity
Keywords: Fullterm Birth; Neonate; Prematurity; Neurodevelopment; Autonomic Nervous System activity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborn: Every child born in the CHU of Saint-Étienne (inborn), any term of its birth, in the hospital neonatal unit at the time of registration (after 37 weeks corrected for prematurity) or in the maternity
  Interventions: Other: Autonomic Nervous System activity

INTERVENTIONS:
Other: Autonomic Nervous System activity — Autonomic activity measured at birth and at 6, 12, 18 and 24 months is represented by time-domain indices (SDNN index, SDANN, pNN50) and frequency- domain indices(PTOT, VLF, LF, HF, ratio LF / HF, LFnu, HFnu), which reflect the short-term variability (parasympathetic branch) and medium term (ortho and parasympathetic branch) of the vegetative balance. This subtle technical assessment of autonomic functioning has been validated in the literature for two decades

SUMMARY:
The heart rate variability assessment of the sympathetic-parasympathetic balance is a strong analytical tool in the autonomic nervous system (ANS) physiology, at each end of life.

In neonatology, it represents an important marker for understanding the breath and cardiac dysfunction, incriminated in the pathophysiology of unexplained death syndrome and apnea-bradycardia of prematurity.

If recent clinical studies conducted by our team highlight a close link between the maturation degree of the ANS and gestational or postnatal age, with a substantial autonomic dysfunction in preterm infants, no study to date has focused profile autonomic maturation in the first two years of life, as that period for the infant is a vulnerability "window" especially cardiopulmonary and neurological.

Psychomotor prognosis of newborns is more serious if prematurity is important and if periventricular leukomalacia or cortical anatomical brain lesions are obvious. However, the conventional imaging (Trans fontanel ultrasound, CT, MRI) is not sufficient in the neonatal period to thoroughly evaluate the neurological risk situations. During the neonatal period, the assessment of autonomic control, in practice easily quantifiable from time and frequency-domain analysis of cardiac RR variability, could be a strong marker, at a given time, from a neurological disorder undetectable by imaging, including sympathetic and parasympathetic nerve conduction dysfunction in some brainstem nuclei and cortical areas.

The postnatal profile of the autonomic balance, as a marker of well ANS regulation could become an additional support to correlate transient or permanent autonomic deficit with a psychomotor development disorder at 2 years of age or later. This tool could be a help to target the children with a neurological risk and to schedule early therapeutic interventions and psychological or educational support.

DETAILED DESCRIPTION:
To meet this objective, we propose to describe for the first time in a cohort of newborns, the cardiac autonomic maturation profile in the first two years of life and the neurological evolution at 2 years.

Main objective.

* Describe the pattern, i.e. the cardiac autonomic maturation during the first two years of life in a cohort of newborns.

Secondary objectives.

* Correlate in this cohort, the autonomous status at birth to the neurological psychomotor status at 2 years.
* Describe the autonomic pattern (evolution profile) during the first two years of life.
* According to specific criteria of pregnancy (maternal smoking, maternal hypertension and gestational age)
* According to data of morphometry (stature and weight development) at birth.
* According to the neonatal morbidity criteria: - bronchopulmonary dysplasia i.e. oxygen dependence at 36 weeks postnatal age, persistent ductus arterious, intra ventricular haemorrhage according to the Papille classification, periventricular leukomalacia, enterocolitis, nosocomial sepsis.
* According to the incidence of serious faintness and rhythmic disorders the two first years of life.

ELIGIBILITY:
Inclusion Criteria:

* Every child born in the CHU of Saint-Étienne (inborn), any term of its birth, in the hospital neonatal unit at the time of registration (after 37 weeks corrected for prematurity) or in the maternity
* Written consent signed by parents
* Parents affiliated in a Social Security regimen

Exclusion Criteria:

* History of intrafamilial dysautonomia
* Heart malformation, congenital abnormality of the brainstem
* Permanent troubles of heart rate
* Any therapy at the time of the study or made in the weeks preceding the study, referred to cardiac or respiratory or known to alter the activity of the ANS
* General anesthesia within 2 weeks prior to registration

Max Age: 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Every child born in the CHU of Saint-Étienne (inborn), any term of its birth, in the hospital neonatal unit at the time of registration (after 37 weeks corrected for prematurity) or in the maternity
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Autonomic activity is represented by time-domain indices and frequency- domain indices, which reflect the short-term variability (parasympathetic branch) and medium term (ortho and parasympathetic branch) of the vegetative balance. | at birth and at 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
the Bayley Scales of Infant Development, developmental with 4 areas of evaluation (motor or postural, oculomotor coordination, language, social relations) to calculate the global and partial quotient Development (QD). | At 24 months
Specific criteria of pregnancy | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Patural H, Teyssier G, Pichot V, Barthelemy JC. [Normal and changed heart rate maturation of the neonate]. Arch Pediatr. 2008 Jun;15(5):614-6. doi: 10.1016/S0929-693X(08)71851-7. No abstract available. French. PMID 18582690
- [Background] Patural H, Pichot V, Jaziri F, Teyssier G, Gaspoz JM, Roche F, Barthelemy JC. Autonomic cardiac control of very preterm newborns: a prolonged dysfunction. Early Hum Dev. 2008 Oct;84(10):681-7. doi: 10.1016/j.earlhumdev.2008.04.010. Epub 2008 Jun 16. PMID 18556151
- [Background] De Rogalski Landrot I, Roche F, Pichot V, Teyssier G, Gaspoz JM, Barthelemy JC, Patural H. Autonomic nervous system activity in premature and full-term infants from theoretical term to 7 years. Auton Neurosci. 2007 Oct 30;136(1-2):105-9. doi: 10.1016/j.autneu.2007.04.008. Epub 2007 Jun 7. PMID 17556047